CLINICAL TRIAL: NCT03956225
Title: Comparison Between iLux and LipiFlow in the Treatment of Meibomian Gland Dysfunction (MGD): A 12-month, Multicenter Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DEG723-P001
Record Dates: First submitted 2019-05-17; First posted 2019-05-20 (Actual); Results first posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Meibomian Gland Dysfunction; Evaporative Dry Eye Disease
Keywords: Dry eye; MGD
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- iLux (Experimental): Single treatment with the Systane iLux Dry Eye System and 12-month follow-up. Both eyes will be treated.
  Interventions: Device: Systane iLux® Dry Eye System
- LipiFlow (Active Comparator): Single treatment with the LipiFlow Thermal Pulsation System and 12-month follow-up. Both eyes will be treated.
  Interventions: Device: LipiFlow® Thermal Pulsation System

INTERVENTIONS:
Device: Systane iLux® Dry Eye System — Commercially available medical device intended for use by qualified eye care professionals to apply localized heat and pressure therapy to a patient's eyelids.
  Arms: iLux
Device: LipiFlow® Thermal Pulsation System — Commercially available medical device intended for use by qualified eye care professionals to apply localized heat and pressure therapy to a patient's eyelids.
  Arms: LipiFlow

SUMMARY:
The purpose of this post-approval study is to demonstrate that iLux treatment offers comparable treatment effectiveness to LipiFlow for MGD treatment at 12 months post single treatment.

DETAILED DESCRIPTION:
Subjects will be expected to attend a total of 8 study visits, including Screening/Baseline, Treatment, and follow-up visits at Week 2 and Months 1, 3, 6, 9, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Understand and sign an Informed Consent document;
* Have Meibomian Gland Dysfunction with evaporative dry eye disease at the screening visit;
* Agree not to wear contact lenses for the duration of the study;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria

* History of eye surgery, as specified in the protocol;
* Eye infection or inflammation, as specified in the protocol;
* Eyelid abnormalities; eyelid tattoos;
* Treated with LipiFlow or iLux in either eye in the last 12 months;
* Contact lens wear within the 1 month prior to Screening;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-10-24 (Actual); Study Completion 2020-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research
Locations (15):
- United States (15):
  - Alcon Investigator 9083, Long Beach, California
  - Alcon Investigator 9081, Los Angeles, California
  - Alcon Investigator 9084, San Diego, California
  - Alcon Investigator 5127, Panama City, Florida
  - Alcon Investigator 4782, Highland Park, Illinois
  - Alcon Investigator 6567, Pittsburg, Kansas
  - Alcon Investigator 5582, Louisville, Kentucky
  - Alcon Investigator 6402, Medina, Minnesota
  - Alcon Investigator 1455, Kansas City, Missouri
  - Alcon Investigator 3828, Poughkeepsie, New York
  - Alcon Investigator 8046, Granville, Ohio
  - Alcon Investigator 6313, Powell, Ohio
  - Alcon Investigator 9082, Chambersburg, Pennsylvania
  - Alcon Investigator 8028, Wichita Falls, Texas
  - Alcon Investigator 5163, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wesley G, Bickle K, Downing J, Fisher B, Greene B, Heinrich C, Kading D, Kannarr S, Miller J, Modi S, Ludwick D, Tauber J, Srinivasan S, Manoj V. Comparison of Two Thermal Pulsation Systems in the Treatment of Meibomian Gland Dysfunction: A Randomized, Multicenter Study. Optom Vis Sci. 2022 Apr 1;99(4):323-332. doi: 10.1097/OPX.0000000000001892. PMID 35383732

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 15 investigative sites located in the United States.
Pre-assignment Details: Of the 299 enrolled subjects, 63 were excluded prior to randomization as screen failures. This reporting group includes all randomized subjects/eyes (236/472).
Units Other Than Participants: eyes
Groups:
- iLux: Single treatment with the Systane iLux Dry Eye System and 12-month follow-up. Both eyes were treated.
- LipiFlow: Single treatment with the LipiFlow Thermal Pulsation System and 12-month follow-up. Both eyes were treated.
Period: Overall Study
Arm/Group | iLux | LipiFlow
Started | 119; 238 eyes | 117; 234 eyes
Completed | 114; 228 eyes | 113; 226 eyes
Not Completed | 5; 10 eyes | 4; 8 eyes
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Other Reasons | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All randomized subjects exposed to any study treatment evaluated in this study
Groups:
- Total: Total of all reporting groups
Arm/Group | iLux | LipiFlow | Total
Number analyzed (Participants) | 119 | 117 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (13.4) | 56.2 (14.1) | 57.3 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 86 | 180
  Male | 25 | 31 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 114 | 115 | 229
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 4 | 10
  White | 103 | 108 | 211
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 119 | 117 | 236

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Change From Baseline in Meibomian Gland Score (MGS) at Month 12
Description: Meibomian glands on the eyelids were assessed by the examiner using a Meibomian Gland Evaluator and a slit lamp microscope. 5 glands in 3 zones (nasal, medial, temporal) were evaluated for each eye and scored from 0 to 3, with a resultant overall score (MGS) of 0 to 45 for each eye. Scoring was follows: 0 = no secretion (worst), 1 = inspissated, 2 = cloudy, 3 = clear liquid (best). A higher change from baseline score indicates an improvement in meibomian gland function.
Time Frame: Baseline, Month 12
Population: Full Analysis Set with data at visit
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | iLux | LipiFlow
Number analyzed (Participants) | 113 | 113
Number analyzed (eyes) | 226 | 226
score on a scale | 17.4 (1.97) | 17.8 (1.98)
Statistical Analysis 1: Comparison: iLux vs LipiFlow; Test type: Non-Inferiority — Noninferiority in change from baseline in MGS was declared if the lower confidence limit (LCL) was greater than -5; Mixed effects repeated measures; Least Squares Mean Difference = -0.3, 95% CI 1-sided [lower limit -2.2], Standard Error of Mean 1.07 — Standard Error of the Least Squares Mean is presented. Least squares mean difference (iLux minus LipiFlow). Lower Confidence Limit is presented

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, up to 12 months.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of participants. This analysis population includes all subjects/eyes exposed to any study treatment evaluated in this study.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study treatment
- iLux Ocular: Events reported in this group occurred in eyes treated with the iLux device
- iLux Nonocular: Events reported in this group occurred in subjects treated with the iLux device
- LipiFlow Ocular: Events reported in this group occurred in eyes treated with the LipiFlow device
- LipiFlow Nonocular: Events reported in this group occurred in subjects treated with the LipiFlow device
Arm/Group | Pretreatment | iLux Ocular | iLux Nonocular | LipiFlow Ocular | LipiFlow Nonocular
All-Cause Mortality (participants affected / at risk) | 0/236 | 0/238 | 0/119 | 0/234 | 0/117
Serious Adverse Events (participants affected / at risk) | 0/236 | 0/238 | 3/119 | 0/234 | 1/117
Other Adverse Events (participants affected / at risk) | 0/236 | 0/238 | 0/119 | 0/234 | 0/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=236) | iLux Ocular (N=238) | iLux Nonocular (N=119) | LipiFlow Ocular (N=234) | LipiFlow Nonocular (N=117)
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
White blood count increased (Investigations) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT03956225/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT03956225/SAP_001.pdf